CLINICAL TRIAL: NCT04751734
Title: Impact of Maternal COVID-19 Vaccination on Breast Milk Antibodies, Milk Bioactive Compounds and Maternal-child Health
Brief Title: Impact of Maternal COVID-19 Vaccines on Breast Milk
Acronym: MilkCorona
Status: Completed | Type: Observational
Sponsor: Institute of Agrochemistry and Food Technology, National Research Council (Other Government)
Collaborators: Hospital Clínico Universitario de Valencia (Other); Hospital Sant Joan de Deu (Other); Hospital Universitario La Fe (Other); Hospital Universitario Doctor Peset (Other); Fundacion Para La Investigacion Hospital La Fe (Other); Universitat Jaume I (Other); University of Barcelona (Other)
Responsible Party: Principal Investigator, Maria Carmen Collado, Researcher, Institute of Agrochemistry and Food Technology, National Research Council
Other Study IDs: IATA-CSIC
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: COVID-19 Vaccines
Keywords: breast milk; microbiota; metabolites; immune compounds; growth and development
MeSH Terms: interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vaccinations: SARS-CoV-2 vaccination
  Interventions: Biological: Covid vaccines

INTERVENTIONS:
Biological: Covid vaccines — women within Priority groups for coronavirus (COVID-19) vaccination

SUMMARY:
prospective multicenter study The main aim is to study the impact of maternal COVID-19 vaccination on breast milk immune, microbiological, and metabolic profile.

ELIGIBILITY:
Inclusion Criteria:

* Priority groups for coronavirus (COVID-19) vaccination (health and social care workers) following breastfeeding practices and receiving vaccines.

Exclusion Criteria:

* cessation of breastfeeding and vaccine side-effects requiring specific treatment and/or hospitalization.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women is Spain
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Antibodies | 1st year
  presence and levels of antibodies

SECONDARY OUTCOMES:
breast milk bioactive composition | 1st year
  immune profile (cytokines and growth factors, immunoglobulins)
breast milk bioactive composition | 1st year
  microbiota profile
breast milk bioactive composition | 1st year
  metabolite profile
infant microbiota | 1st year
  infant microbiota composition and diversity
infant growth and development | 1st year
  z-scores growth curves

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Fundacion Investigacion Sanitaria INCLIVA, Valencia
  - Hospital Universitario y Politecnico la Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Selma-Royo M, Bauerl C, Mena-Tudela D, Aguilar-Camprubi L, Perez-Cano FJ, Parra-Llorca A, Lerin C, Martinez-Costa C, Collado MC. Anti-SARS-CoV-2 IgA and IgG in human milk after vaccination is dependent on vaccine type and previous SARS-CoV-2 exposure: a longitudinal study. Genome Med. 2022 Apr 21;14(1):42. doi: 10.1186/s13073-022-01043-9. PMID 35449030